CLINICAL TRIAL: NCT00513669
Title: A Phase Ib Double-blind Randomized Placebo Controlled Age-deescalating Trial of Two Virosome Formulated Anti-malaria Vaccine Components (PEV 301 and PEV 302) Administered in Combination to Healthy Semi-immune Tanzanian Volunteers
Brief Title: Phase Ib Trial of Two Virosome Formulated Malaria Vaccine Components (PEV 301, PEV 302) in Tanzania
Acronym: PMAL03
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Mymetics Corporation (Industry); Pevion Biotech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PMAL03
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Falciparum Malaria
Keywords: Malaria; Vaccine; Falciparum; Trial; Phase I; Safety; Immunogenicity
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Virosomes; Inflexal V

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 PEV301&302 (Experimental): The vaccine includes two antigens (CSP and AMA1- derived)in combination and formulated with virosomes
  Interventions: Biological: PEV 301& 302 in virosomes
- 2 Influenza vaccine (Active Comparator): Inflexal V is the comparator that includes 3 antigens from flu formulated in virosomes
  Interventions: Biological: Inflexal V (active comparator)

INTERVENTIONS:
Biological: PEV 301& 302 in virosomes — PEV 301 50 µg plus PEV 302 10 µg formulated in virosomes and injected at day 0 and 90
  Arms: 1 PEV301&302
Biological: Inflexal V (active comparator) — Inflexal V is a marketed influenza vaccine that will be given at day 0 and 90
  Arms: 2 Influenza vaccine

SUMMARY:
This is a phase Ib double-blind randomized placebo controlled age-deescalating trial to assess sagety and immunogenicity of two virosome formulated anti-malaria vaccine components (PEV 301 and PEV 302) administered in combination to healthy semi-immune Tanzanian adult and children.

DETAILED DESCRIPTION:
Volunteers will be screened, enrolled, injected with the vaccine or comparator and followed by the clinicians at the Bagamoyo Research and Training Unit of the the Ifakara Health Research and Development Center (BRTU-IHRDC).

First, 10 adult males will be enrolled and randomized in 2 groups: Group AV (n=8) will be injected with the vaccine combination and group AP (n=2) will be vaccinated with the placebo=comparator (Inflexal V). 5 weeks later, 8 children will be enrolled first and randomized in 2 groups: Group CV (n=6) will be injected with the vaccine combination and group CP (n=2) will be vaccinated with comparator. 1 week later, the rest of the cohort (n=32) will be enrolled and randomized in 2 groups: Group CV (n=26) will be injected with the vaccine combination and group CP (n=6) will be vaccinated with comparator.

Immunogenicity assessments for humoral immune response will be made at baseline (days -10 to -2), day 30 (+4), day 90 (+4) (day of 2nd vaccination), 120 (+4), 180 (+7), and 365 (+14).

Cellular immune responses will be assessed before 1st vaccination (day 0), two weeks after 2nd vaccination (day 104 ±2), and one year after the 1st vaccination (day 365) Safety assessments will be made by the investigator at baseline (days -10 to -2, before the 1st immunization) and at day 1, 2, 3, 7, 14, 30 after each vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Male volunteers aged between 18 and 45 years for the adult group, and children of both sexes aged 5-9 years for schoolchildren group
2. Written informed consent obtained from the volunteer (adult) or guardian/ legal representative (children). In case patient is illiterate, an impartial witness should be present during the entire consent procedure
3. Free of obvious health problems as established by medical history and clinical examination before entering the study
4. Body Mass Index between 18 and 30 for adults; MUAC less than 12 for children

Exclusion Criteria:

1. Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period and safety follow-up
2. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose
3. Any chronic drug therapy to be continued during the study period
4. Any confirmed or suspected acquired immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection, or history of congenital or hereditary immunodeficiency
5. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
6. Acute disease at the time of enrollment. Acute disease is defined as the presence of a moderate or severe illness with or without fever (defined as temperature more than 37.5°C)
7. Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests
8. Acute or chronic diabetes
9. History of chronic alcohol consumption and/or intravenous drug abuse

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety (incidence of local and systemic adverse events) Humoral immunity | 30 days post-injection

SECONDARY OUTCOMES:
Cell-mediated immunity | 14 days post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Blaise Genton, MD PhD, Principal Investigator — Swiss tropical institute, Ifakara Health Research and Development Center
Locations (1):
- Bagamoyo Research and Training Unit, Bagamoyo, Tanzania

REFERENCES:
- [Derived] Cech PG, Aebi T, Abdallah MS, Mpina M, Machunda EB, Westerfeld N, Stoffel SA, Zurbriggen R, Pluschke G, Tanner M, Daubenberger C, Genton B, Abdulla S. Virosome-formulated Plasmodium falciparum AMA-1 & CSP derived peptides as malaria vaccine: randomized phase 1b trial in semi-immune adults & children. PLoS One. 2011;6(7):e22273. doi: 10.1371/journal.pone.0022273. Epub 2011 Jul 22. PMID 21799810
- See also: Website of the Swiss Tropical Institute — http://www.sti.ch